CLINICAL TRIAL: NCT02950948
Title: Prospective, Randomised, Double-blind, Placebo Controlled, Phase III Clinical Study Assessing the Efficacy of 25 mg Natural Progesterone Administered Subcutaneously in Restoring the Normal Luteal Phase in Women With Previous Diagnosis of Luteal Phase Deficiency
Brief Title: Progesterone in Luteal Phase Deficiency
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: inability to recruit an adequate number of subjects.
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16I-Prg05
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Luteal Phase Defect
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progesterone (Experimental): 25 mg of progesterone will be administered daily by subcutaneous injection.
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): 25 mg of progesterone will be administered daily by subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — Progesterone will be administered subcutaneously once a day for 14 days/month, for 12 months.
  Other Names: Test
  Arms: Progesterone
Drug: Placebo — A placebo solution will be administered subcutaneously once a day for 14 days/month, for 12 months.
  Other Names: Control
  Arms: Placebo

SUMMARY:
The main objective of this study will be to assess the efficacy of natural progesterone at a daily dose of 25 mg in restoring a normal luteal phase. The primary end-point will be the ongoing pregnancy rate.

The secondary objectives will be the rate of endometrial biopsy showing an in phase endometrium after 3 months of treatment.

The length of the luteal phase of the menstrual cycle after treatment will also be assessed and compared with the initial duration (from LH peak to onset of menstruation).

ELIGIBILITY:
Inclusion Criteria:

* Women who wish to get pregnant with a previous diagnosis of luteal phase deficiency:
* Able and willing to sign the Subject Consent Form and adhere to the study visit schedule;
* Age: 20-35 years;
* BMI: 18-28 kg/m2;
* Inadequate luteal phase (menstrual period shorter than 21 days);
* Sub-fertile couple: 12 months of trying to conceive without success.
* Normal uterine cavity;
* Basal P4 level (day 3 of a previous cycle) ≤ 3ng/ml;
* Non-smoking;
* Fertile male partner (normal sperm count).

Exclusion Criteria:

* History of recurrent miscarriage;
* Basal P4 level (day 3 of a previous cycle) > 3ng/ml;
* Severe uterine malformations (including submucosal fibroids, endometrial polyps, and intrauterine adhesions) ;
* Known hypersensitivity to study medication;
* Neoplasias (known or suspected breast or genital tract cancer);
* Severe impairment of hepatic or renal function;
* Use of concomitant medications that might interfere with study evaluations (other hormonal treatment);
* Current vaginal infection;
* Endometriosis;
* PCOS;
* Partially or completed block of fallopian tubes;
* Hydrosalpinx;
* Active arterial or venous thromboembolism or severe thrombophlebitis, or a history of these events;
* Porphyria;
* A history of idiopathic jaundice, severe pruritus or pemphigoid gestationis during pregnancy;
* Antiphospholipid syndrome;
* Diabetes mellitus;
* Thyroid diseases or autoimmune conditions;
* Hypothalamic dysfunction;
* Hyperprolactinaemia;
* Infertility due to male factor;
* Smokers.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate at 12 weeks of gestation | 12 weeks

SECONDARY OUTCOMES:
Rate of in phase endometrial biopsies | 3 months
Length of luteal phase | 3 months